CLINICAL TRIAL: NCT00002503
Title: A PROSPECTIVE MULTICENTER RANDOMIZED STUDY COMPARING STRONTIUM-89 CHLORIDE AND PALLIATIVE LOCAL FIELD RADIOTHERAPY IN PATIENTS WITH HORMONAL ESCAPED ADVANCED PROSTATIC CANCER
Brief Title: Strontium Compared With Radiation Therapy in Treating Patients With Hormone-Refractory Prostate Cancer With Painful Bone Metastases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-30921; EORTC-30921
Record Dates: First submitted 1999-11-01; First posted 2004-05-20 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Metastatic Cancer; Prostate Cancer
Keywords: recurrent prostate cancer; bone metastases
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — strontium chloride

INTERVENTIONS:
Radiation: strontium chloride Sr 89

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. This may be an effective treatment for prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of strontium or radiation therapy in treating patients with prostate cancer that is refractory to hormone therapy who have painful bone metastases.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare, in a randomized Phase III setting, the subjective response rate, time to progression, and survival of patients with hormone-refractory prostate cancer with painful osseous metastases treated with either strontium-89 or palliative local radiotherapy. II. Compare the quality of life achieved on these two regimens. III. Determine the toxicity and morbidity of treatment on these two regimens. IV. Compare the cost effectiveness of these two regimens.

OUTLINE: Randomized study. Arm I: Radioisotope therapy. Strontium-89 chloride, Strontium-89. Arm II: Radiotherapy. Involved-field irradiation (equipment unspecified).

PROJECTED ACCRUAL: 200 patients will be entered over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven carcinoma of the prostate that has relapsed subsequent to chemical or surgical castration and/or antiandrogen therapy Painful, unirradiated osseous metastasis required Documentation by bone scan and x-ray required Number and extent of metastases determined according to Soloway and fitting grades 1-3 Prior hormonal therapy must have lasted at least 3 months and must be continued until completion of this study No imminent paraplegia related to metastases No uncorrectable urinary incontinence

PATIENT CHARACTERISTICS: Age: Any age Performance status: WHO 0-2 Hematopoietic: WBC greater than 3,500 Platelets greater than 150,000 Hepatic: Not specified Renal: Creatinine no greater than 2.2 mg/dl (200 micromoles/liter) Other: No calcium supplementation No second malignancy except basal cell skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No restriction Endocrine therapy: Prior and concurrent hormonal therapy required Radiotherapy: No prior strontium-89 No prior hemibody or total-body irradiation Prior local-field irradiation for bone metastases allowed provided new site of painful metastases exists Surgery: Surgical castration allowed

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 1992-10; Primary Completion 2000-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: G. O. N. Oosterhof, MD, PhD, Study Chair — Academisch Ziekenhuis Maastricht
Locations (21):
- Belgium (4):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - U.Z. Gasthuisberg, Leuven
- Denmark (2):
  - Aarhus Kommunehospital, Aarhus
  - Rigshospitalet, Copenhagen
- Italy (5):
  - Ospedale B. Ramazzini, Carpi
  - Universita Degli Studi di Firenze - Policlin. di Careggi, Florence
  - Instituto Scientifico H.S. Raffaele, Milan
  - San Raffaele Hospital, Rome
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Netherlands (5):
  - Groot Ziekengasthuis 's-Hertogenbosch, 's-Hertogenbosch
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - University Medical Center Nijmegen, Nijmegen
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
- Hospital Santa Maria, Lisbon, Portugal
- Medical Radiological Research Center, Obninsk, Russia
- Inselspital, Bern, Bern, Switzerland
- Newcastle General Hospital, Newcastle upon Tyne, England, United Kingdom

REFERENCES:
- [Result] Oosterhof GO, Roberts JT, de Reijke TM, Engelholm SA, Horenblas S, von der Maase H, Neymark N, Debois M, Collette L. Strontium(89) chloride versus palliative local field radiotherapy in patients with hormonal escaped prostate cancer: a phase III study of the European Organisation for Research and Treatment of Cancer, Genitourinary Group. Eur Urol. 2003 Nov;44(5):519-26. doi: 10.1016/s0302-2838(03)00364-6. PMID 14572748